CLINICAL TRIAL: NCT06488118
Title: Lung Immune Challenge Study Controlled Exposure to Inhaled Resiquimod (R848) to Study Mechanisms of Inflammation
Brief Title: Lung Immune Challenge Study: Controlled Exposure to Inhaled Resiquimod (R848)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akhilesh Jha (Other)
Collaborators: University of Cambridge (Other)
Responsible Party: Sponsor-Investigator, Akhilesh Jha, MRC Clinician Scientist, Cambridge University Hospitals NHS Foundation Trust
Organization: Cambridge University Hospitals NHS Foundation Trust (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: A096886; MR/Y000935/1 (Other Grant/Funding Number: Medical Research Council (MRC))
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Innate Immunity; Mucosal Immunity; Asthma; Viral Infection
Keywords: Asthma; Immunology; Viral infection; Airway Epithelium; Respiratory Medicine; Innate Immunity; Sputum
MeSH Terms: conditions — Asthma; Virus Diseases | interventions — resiquimod; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- R848 0.1 μg/mL (Active Comparator): Inhaled Resiquimod (R848) 0.1 μg/mL
  Interventions: Drug: R848
- R848 1.0 μg/mL (Active Comparator): Inhaled Resiquimod (R848) 1.0 μg/mL
  Interventions: Drug: R848
- R848 10 μg/mL (Active Comparator): Inhaled Resiquimod (R848) 10 μg/mL
  Interventions: Drug: R848
- R848 100 μg/mL (Active Comparator): Inhaled Resiquimod (R848) 100 μg/mL
  Interventions: Drug: R848
- Saline (Placebo Comparator): Inhaled Saline
  Interventions: Drug: Saline
- Asthma volunteers inhaled R848 (Active Comparator): Highest tolerated dose inhaled R848 in healthy volunteers to be given to volunteers with asthma
  Interventions: Drug: R848
- Asthma volunteers inhaled saline (Placebo Comparator): Inhaled saline to be given to volunteers with asthma
  Interventions: Drug: Saline
- Sample only (No Intervention): Sample only collection from volunteers for protocol optimisation

INTERVENTIONS:
Drug: R848 — Inhaled R848 dose ranging from 0.1 to 100 μg/mL
  Arms: Asthma volunteers inhaled R848; R848 0.1 μg/mL; R848 1.0 μg/mL; R848 10 μg/mL; R848 100 μg/mL
Drug: Saline — Inhaled Saline control
  Arms: Asthma volunteers inhaled saline; Saline

SUMMARY:
Respiratory viral infections can be a cause of significant illness, particularly in vulnerable individuals as seen in the COVID-19 pandemic. An underactive or overactive immune response can lead to ineffective resolution of inflammation after an infection, especially in people with airway diseases such as asthma. A better understanding of immune responses to infection that does not rely on cell or animal models is crucial to help develop better treatments for lung inflammation.

An established method of studying inflammation in humans is through careful and controlled exposure (or "challenge") with a mimic of a virus to simulate an infection in a similar manner to that of a virus, but with the advantage of not causing an infection. The investigators have already developed a well-tolerated mimic of human viral infection using a sterile substance called Resiquimod (or R848). Since it does not contain living organisms there is no possibility of being infected. This has been used previously as a nasal spray to cause a mild short-lived inflammation that mimics a mild cold. This has been used safely in a range of people of different ages including those who have asthma.

There are differences however in how the nose and lungs respond to viral infections. This is particularly true in those with airway diseases such as asthma, who have cells in the airways of their lungs that respond in a different way to inflammatory triggers (such as viruses).

The current study aims to build on previous research by developing a new approach of studying inflammation in the lungs using a small volume of Resiquimod. This will be done by gently inhaling a fine mist through a mouthpiece into the lungs. Blood and phlegm samples would then be collected to assess inflammation and how well people tolerate the procedure.

DETAILED DESCRIPTION:
Background The initial immune response to respiratory viral infections is key to determining what kind of clinical outcome is experienced. The COVID-19 pandemic highlights the key importance of gaining a thorough understanding of these immune mechanisms.

People with chronic lung conditions such as asthma often experience more severe and prolonged symptoms in response to external triggers. This can be due to ongoing inflammation in their airways and lungs. Animal and cell models fail to accurately recapitulate the disease, which limit its usefulness in developing new treatments.

Observational human studies of asthma attacks can be useful but have several confounding factors, which significantly influence the outcomes being assessed. For example, one issue may be the significant variability in time between exposure to a pathogen to the point at which they present to hospital.

One important method for understanding mechanisms of inflammation in humans, is to perform controlled and careful exposure to an inflammatory stimulus to assess why and how differences occur between individuals. This is already established using live viral infection studies - however these studies are technically difficult, resource intensive, may make participants feel unwell for several days, and can be inconvenient for them due to the need for prolonged quarantine.

An alternative approach for studying the first line of immune defence (or "innate immunity"), is to use a mimic of a virus that binds to the same receptors as respiratory viruses such as influenza and SARS-CoV-2. The study team have already established and published this research using a nasal spray with a synthetic compound called Resiquimod (R848). It generates an inflammatory response with the release of molecules such as interferons and cytokines in the nose in a very similar manner to what we see with live viral infections. This approach has been used to demonstrate differences in immune responses between healthy individuals and people with asthma.

However, there are important differences between how the nose and lungs may respond to an inflammatory stimulus. This is due to many reasons including differences in the types of cells present between the upper and lower airways, which is especially the case in people who have airway diseases such as asthma.

Lung Challenge Model A lung immune challenge model using Resiquimod would therefore represent an important approach for studying differences in innate immune responses between individuals, enable an understanding of which cells are responsible for driving inflammation, and have the potential to be a platform for testing new anti-inflammatory therapies.

The first step of this approach and the focus of the current study is to define what dose is the most suitable for generating an appropriate innate immune response, whilst also being clinically tolerable for volunteers. The dose has already been established in the respiratory tract using nasal challenge, so this is a very good starting point when designing the current study. The initial dose for lung challenge will be 100-fold lower than with nasal challenge and therefore it is not anticipated to generate an immune response. The subsequent doses will then be escalated and reach a maximum dose that has already been administered via the intranasal route in clinical trials.

Identifying whether an appropriate immune response has been generated will be done by measuring the inflammatory molecule CXCL10. It is known that CXCL10 is an excellent biomarker for immune activation as it is increased after nasal challenge with Resiquimod, as well as after natural viral infections. CXCL10 will be measured in the blood and in the lungs by analysing sputum samples.

The dose cohort design with 6 participants in each dose cohort, and 4 participants being randomised to Resiquimod, whilst 2 participants being randomised to saline is based on an already published AstraZeneca trial of a similar compound used for inhaled challenge. This will enable an accurate comparison of responses between saline and active groups.

An important aspect of this study is to ensure it is clinically tolerable for volunteers. They will have been informed in the PIS that they may experience flu-like symptoms as the purpose of the study is to mimic flu and therefore, they may have transient inflammation and cold symptoms. To ensure their safety - their symptoms, physiological observations, and airway function will be closely monitored for the first 24 hours of the study directly within the research facility with access to full healthcare resources and staff. Individuals with asthma will only undergo inhaled challenge once an appropriate dose has been established in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged between 18 and 60 years.
* Willing and able to give informed consent for participation in the study.
* Female participants of child-bearing potential and male participants whose partner is of child-bearing potential must be willing to ensure that they or their partner use effective contraception during the study.
* Clinically acceptable laboratory measurements and ECG at enrolment.
* Ability to expectorate sputum.
* Optional additional swab for SARS-CoV-2 testing will be collected from participants if required by local or/and national health and safety policies at the time of sampling.

For healthy volunteers:

* No clinical history of asthma
* Normal baseline spirometry i.e. FEV1/Forced Vital Capacity (FVC) ratio z-score greater than the lower limit of normal.

For volunteers with asthma:

* Physician-diagnosed mild to moderate asthma which is not poorly controlled as evidenced by an Asthma Control Questionnaire (ACQ-5) score of ≤1.5.
* They are permitted to be on inhaled corticosteroids (ICS), long-acting beta agonist (LABA) and long-acting muscarinic antagonists (LAMA).
* Pre-bronchodilator FEV1 ≥70% predicted.
* Evidence of bronchial hyperreactivity as evidenced by either (i) Bronchodilator reversibility (increase FEV1 ≥12% and 200 mL); (ii) Positive methacholine challenge (PC20 < 8mg/ml), or (iii) Positive challenge test as per current CUH policy.

Exclusion Criteria:

* Upper respiratory tract infection in preceding 14 days.
* Lower respiratory tract infection in preceding 28 days.
* Female participants who are pregnant, lactating or planning pregnancy.
* Respiratory diseases (other than asthma where specified).
* Significant extrapulmonary medical conditions.
* Extreme obesity (BMI >40).
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational product in the past 12 weeks.
* No newly prescribed courses of medication including corticosteroids in the four weeks before first study dose other than mild analgesia, vitamins, and supplements.
* Smoking tobacco or vaping products in previous 6 months.
* Smoking history of >5 pack years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male (Cisgender) Female (Cisgender)
Enrollment: 36 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in Serum or Sputum CXCL10 | 3 weeks from screening visit until 24 hours after inhaled R848 challenge
  Change in CXCL10 in serum or induced sputum before and after inhaled R848

SECONDARY OUTCOMES:
Change in FEV1 | Change in FEV1 at 1, 4, 8, 24 and 48 hours after single ascending dose inhaled R848 or saline
  Change in FEV1 after single ascending dose inhaled R848 or saline
Change in Temperature | Change in temperature (degrees celsius) at 1, 4, 8, 24 and 48 hours after single ascending dose inhaled R848 or saline
  Change in temperature (degrees celsius) after single ascending dose inhaled R848 or saline
Change in Pulse Rate | Change in Pulse Rate at 1, 4, 8, 24 and 48 hours after single ascending dose inhaled R848 or saline
  Change in Pulse Rate after single ascending dose inhaled R848 or saline
Change in Systolic Blood Pressure | Change in systolic blood pressure at 1, 4, 8, 24 and 48 hours after single ascending dose inhaled R848 or saline
  Change in systolic blood pressure after single ascending dose inhaled R848 or saline
Change in Peripheral Eosinophil Counts | Change in peripheral eosinophil counts at 4, 24 and 48 hours after single ascending dose inhaled R848 or saline
  Change in peripheral eosinophil counts after single ascending dose inhaled R848 or saline
Change in Peripheral Lymphocyte Counts | Change in peripheral lymphocyte counts at 4, 24 and 48 hours after single ascending dose inhaled R848 or saline
  Change in peripheral lymphocyte counts after single ascending dose inhaled R848 or saline
Change in Serum CRP | Change in serum CRP at 4, 24 and 48 hours after single ascending dose inhaled R848 or saline
  Change in serum CRP after single ascending dose inhaled R848 or saline

CONTACTS AND LOCATIONS:
Locations (1):
- NIHR Cambridge Clinical Research Facility, Cambridge, Cambridgeshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jha A, Thwaites RS, Tunstall T, Kon OM, Shattock RJ, Hansel TT, Openshaw PJM. Increased nasal mucosal interferon and CCL13 response to a TLR7/8 agonist in asthma and allergic rhinitis. J Allergy Clin Immunol. 2021 Feb;147(2):694-703.e12. doi: 10.1016/j.jaci.2020.07.012. Epub 2020 Jul 24. PMID 32717253
- [Background] Progatzky F, Jha A, Wane M, Thwaites RS, Makris S, Shattock RJ, Johansson C, Openshaw PJ, Bugeon L, Hansel TT, Dallman MJ. Induction of innate cytokine responses by respiratory mucosal challenge with R848 in zebrafish, mice, and humans. J Allergy Clin Immunol. 2019 Jul;144(1):342-345.e7. doi: 10.1016/j.jaci.2019.04.003. Epub 2019 Apr 16. No abstract available. PMID 31002833
- See also: Study website — https://lungchallenge.org.uk/

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-14): https://cdn.clinicaltrials.gov/large-docs/18/NCT06488118/Prot_SAP_000.pdf
  • Informed Consent Form (2024-04-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT06488118/ICF_001.pdf